CLINICAL TRIAL: NCT04501510
Title: The Use of Ultrasonography as a Diagnostic Tool for the Fracture Management
Brief Title: Ultrasonography in Fracture Management
Acronym: UFrac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Anna Malwina Kamelska-Sadowska, PhD, University of Warmia and Mazury
Other Study IDs: 61.610.022-110
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Fractures, Bone; Upper Extremity Injury; Healing Fracture of Bone; Vascularization
Keywords: ultrasonography; bone; fracture; x-ray; injury; upper extremity; humerus; radius; vascularization; Doppler
MeSH Terms: conditions — Fractures, Bone; Arm Injuries; Neovascularization, Pathologic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HumerusFracture: Patients with humerus fracture
  Interventions: Diagnostic Test: Ultrasonographic examination validation and testing
- RadiusFracture: Patients with radial bone fracture
  Interventions: Diagnostic Test: Ultrasonographic examination validation and testing

INTERVENTIONS:
Diagnostic Test: Ultrasonographic examination validation and testing — X-ray imaging as well as the ultrasonographic examination of the fracture and healing process in children will be performed. The validation of an usg will be done.

SUMMARY:
The bone fracture is usually diagnosed using an X-ray examination (the method of choice). However, in the case of the youngest patients (children and adolescents), it carries a potential risk of X-ray radiation exposure. What is important, an X-ray examination often fails to detect occult fractures or the early stages of a fracture with or without bone fusion. The literature emphasizes that from 2 to 36% of fractures may be unnoticed on X-ray images (false negative results). Therefore, additional possibilities are sought to improve the initial diagnosis.

It was shown that ultrasound could be used instead of the conventional imaging. The most important advantages of the usg are the absence of radiation exposure and greater availability. Moreover, the evaluator is able to show neovascularization during usg examination, which is important in bone healing process.

The aim of this study is (1) to validate the ultrasound imaging method for the fracture management; (2) to use an ultrasound imaging to assess the bone fracture and healing process during 8 weeks post injury.

This study consists of 50 patients aged 10-18 years old. The forearm fracture will be diagnosed using an X-ray imaging as well as an ultrasound imaging in the first 3 days post injury (initial study). It is planned to assess the healing process after 2, 4, 6 and/or 8 weeks post injury (comparative study).

DETAILED DESCRIPTION:
The physiological fracture healing is based on the proper facilitation of regeneration and proliferation process. The bone fracture is usually diagnosed using an X-ray examination. However, an ultrasound imaging could be used instead of the conventional imaging. It is important in the case of the youngest patients. In these cases, the Hubner protocol/algorithm is often used. The patients with suspected fracture are advised to perform an ultrasound examination. Only after the confirmation of a suspected fracture, an X-ray examination should be performed.

Bone structure show typical characteristics, which make an ultrasonography an attractive medical diagnostic tool. Highly dense tissues such as bone reflect echoes and, therefore, appear bright white on an ultrasound (reflection from the cortical surface of the bone). This allows bone to be clearly distinguished from the surrounding soft tissues.

It was shown that ultrasound is a good diagnostic tool to assess the fracture healing process. The advantage of usg is that it is non-invasive, does not use ionizing radiation and is performed in a real-time.

The first study about the ultrasound in the diagnosis of fracture was carried out in 1988 in a group of 41 newborns with suspected clavicle fractures after complicated delivery. In all cases, the collarbone fracture was easily identifiable by an ultrasound in the first few days after the injury. Moreover, these data correlated with the conventional X-ray imaging.

It was also shown that the ultrasound method in pediatric patients can be used to visualize fractures, e.g. of the ribs or the sternum. In the acute phase, disturbances in the cortical layer of the bone as well as recent hematoma are easily observed. In the later phase, the formation of a callus (callus hypertrophy) could be diagnosed.

The aim of this study is (1) to validate the ultrasound imaging method using variables such as repeatability, interclass correlation coefficient (Qw), relative standard deviation (rSD) etc.; (2) to use an ultrasound imaging to assess the bone fracture and healing process during 8 weeks post injury.

This study consists of 50 patients aged 10-18 years old. The forearm fracture will be diagnosed using an X-ray imaging as well as an ultrasound imaging in the first 3 days post injury (initial study). It is planned to assess the proper healing process after 2, 4, 6 and/or 8 weeks post injury (comparative study).

Ultrasound examination:

* the measurement of the humerus in two different projections (a-p and lateral). The distance from the acromion localized on the shoulder blade will be measured in order to repeat the examination in the same area.
* radial bone examination in two different projections (a-p and lateral). The distance from the radiocarpal joint space will be measured in order to repeat the examination in the same area.
* additionally, POWER Doppler assessment of callus neovascularization will be performed (each recording of the Doppler frame parameters for a given patient in order to repeat the examination at subsequent controls)

Experimental Design:

The fracture diagnosis is planned to be performed on the day of the injury, or at an interval of no more than 2-3 days post the injury as an initial examination and approx. during 8 weeks after the injury as a comparative examination (during the first control in an orthopedic clinic after 14 days, 4 weeks, 6 weeks and/or 8 weeks).

All the procedures performed in this study involving human participants will conform to the ethical guidelines of the 1975 Declaration of Helsinki (and its later amendments or comparable ethical standards, revised in 2013) and follow the Adapted Physical Activity (APA) Ethics Standard.

The protocol was approved by the Ethics Committee of Stanislaw Popowski Regional Specialized Children's Hospital in Olsztyn, Poland (number of approval: 6 ZE//2020/WSSD; date of approval: 22 May 2020).

The experiment will be conducted with the understanding of each subject. All subjects as well as their parents will give written informed consent before children's participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* the proximal end of the humerus and the distal end of the radius bones fractures
* voluntary participation and consent to participate in the study signed by the parent and patient
* declaration of participation in an X-ray and ultrasound examination during all 8 weeks post-injury
* no medical contraindications to participate in the study program

Exclusion Criteria:

* previous injuries of a similar body area
* plaster immobilization
* fractures referred for surgery

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 50 patients admitted to the Orhopaedics and Trauma Ward of Prof. dr Stanislaw Popowski Regional Specialized Children's Hospital in Olsztyn, Poland with trauma to the upper extremity (from the proximal of the wrist to distal of the glenohumeral joint with evidence of pain, tenderness or swelling of the limb). Patients will be devided into two groups of radius or humerus bone (RadiusFracture and HumerusFracture groups). All patients will be recruited starting from July 2020. In all patients, first ultrasound and then standard plain radiography will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in fracture management using x-ray imaging and medical ultrasound within 8 weeks post-injury | through study completion, an average of 1 year
  The confirmation of fracture and healing process
Mean Change from Baseline in adhesions development using medical ultrasound within 8 weeks post-injury | through study completion, an average of 1 year
  The assessment of the development of adhesions (changes in soft tissue image)
Mean Change from Baseline in vascularization on POWER Doppler within 8 weeks post-injury | through study completion, an average of 1 year
  Mean Change from Baseline in vascularization on POWER Doppler within 8 weeks post-injury
Mean Change from Baseline in Pain Scores on the Visual Analog Scale within 8 weeks post-injury | through study completion, an average of 1 year
  The changes in pain scale will be assessed using Visual Analogue Scale (VAS) and other specific for the selected injuries. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' (from mild to severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Kamelska-Sadowska, PhD, Study Chair — Department of Rehabilitation and Orthopedics, Collegium Medicum, Faculty of Medicine, University of Warmia and Mazury in Olsztyn
Locations (1):
- University of Warmia and Mazury in Olsztyn, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maffulli N, Hughes T, Fixsen JA. Ultrasonographic monitoring of limb lengthening. J Bone Joint Surg Br. 1992 Jan;74(1):130-2. doi: 10.1302/0301-620X.74B1.1732241.
- [Background] Cho KH, Lee SM, Lee YH, Suh KJ. Ultrasound diagnosis of either an occult or missed fracture of an extremity in pediatric-aged children. Korean J Radiol. 2010 Jan-Feb;11(1):84-94. doi: 10.3348/kjr.2010.11.1.84. Epub 2009 Dec 28. PMID 20046499
- [Background] Malahias MA, Manolopoulos PP, Kadu V, Shahpari O, Fagkrezos D, Kaseta MK. Bedside Ultrasonography for Early Diagnosis of Occult Radial Head Fractures in Emergency Room: A CT-Comparative Diagnostic Study. Arch Bone Jt Surg. 2018 Nov;6(6):539-546. PMID 30637310
- [Background] Hubner U, Schlicht W, Outzen S, Barthel M, Halsband H. Ultrasound in the diagnosis of fractures in children. J Bone Joint Surg Br. 2000 Nov;82(8):1170-3. doi: 10.1302/0301-620x.82b8.10087. PMID 11132281
- See also: Erik Beek and Rick R van Rijn (eds). Diagnostic Pediatric Ultrasound — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5105360/